CLINICAL TRIAL: NCT00103974
Title: A Phase I Trial of Immunotherapy With BHT-3009 Alone or Combined With Atorvastatin in Patients With Multiple Sclerosis
Brief Title: Immunotherapy With BHT-3009 Alone or Combined With Atorvastatin in Patients With Multiple Sclerosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayhill Therapeutics (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: BHT-3009-01
Record Dates: First submitted 2005-02-17; First posted 2005-02-18 (Estimated); Last update posted 2008-04-07 (Estimated); Status verified 2008-02

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; relapsing-remitting; secondary progressive
MeSH Terms: conditions — Multiple Sclerosis

INTERVENTIONS:
Biological: BHT-3009-01

SUMMARY:
This research study is being done to evaluate the safety of BHT-3009 alone and when combined with atorvastatin (Lipitor) in patients with multiple sclerosis (MS).

DETAILED DESCRIPTION:
This research study is being done to evaluate the safety of BHT-3009 alone and when combined with atorvastatin (Lipitor) in patients with multiple sclerosis (MS).

Patients with MS are thought to have an immune response that attacks certain proteins in the brain, including myelin basic protein. (Myelin basic protein is a protein that makes up part of the outside layer of nerve cells.) BHT-3009 is an investigational immunotherapy product that is designed to alter the immune response to myelin basic protein and make the response less harmful. BHT-3009 contains the DNA (gene) for myelin basic protein.

Three different doses of BHT-3009 will be tested to determine if there are any differences in safety or effects on immunity. This is the first clinical research study of BHT-3009. Laboratory studies have shown that BHT-3009 and atorvastatin given together alters the immune response to myelin basic protein and makes the response less harmful.

ELIGIBILITY:
Inclusion Criteria:

* Definite diagnosis of multiple sclerosis by the McDonald criteria.
* Patients with relapsing remitting MS or secondary progressive MS are eligible.
* 1-5 gadolinium enhancing (Gd+) lesions on the first Screening MRI or relapse in the previous 2 years, or disease worsening in the previous 2 years
* Clinically stable for > 1 month before screening evaluation and during screening. Patients who are stable on approved therapy are eligible only if they have intolerable side effects or other medical reasons for discontinuing approved therapy.
* Off interferon for > 1 month before screening evaluation.
* Off immunosuppressive and cytotoxic therapy (e.g. mitoxantrone, cladrabine) >12 months or > 6 months with CD4 count > 400.
* EDSS ≥ 2.5 and < 7.0.
* Female or male, age > 18 years.
* Able to give informed consent.
* WBC and platelets in normal range, hemoglobin > 10.0 g/dl.
* AST, ALT, bilirubin < upper limit of normal.
* Creatinine < upper limit of normal.
* CPK < upper limit of normal.

Exclusion Criteria:

* High-dose corticosteroids (e.g. >500 mg methylprednisolone or equivalent) within previous month.
* >5 Gd+ lesions on the first Screening MRI.
* Previous vaccine therapy, stem cell transplantation or total lymphoid radiation.
* Glatiramer within previous 12 months.
* Treatment with any statin in the previous 6 months or elevated cholesterol that requires treatment with a statin.
* Pregnant or lactating women.
* Unwilling to use a medically acceptable form of birth control.
* History of positive test for HIV, hepatitis B or hepatitis C.
* Clinically significant ECG abnormalities.
* Medical condition or social circumstances that would in the opinion of the investigator prevent full participation in the trial or evaluation of study endpoints.
* Implanted pacemakers, defibrillators or other metallic objects on or inside the body that limit performing MRI scans.
* History of intolerable adverse events with statin therapy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2004-07; Study Completion 2007-03

PRIMARY OUTCOMES:
Evaluate safety of BHT-3009 alone and when combined with atorvastatin in patients with multiple sclerosis.
Determine dose of BHT-3009 and regimen for phase II testing.

SECONDARY OUTCOMES:
Describe effect of treatment on antibody and T cell responses to myelin basic protein (MBP).
Describe clinical course of treated patients.
Explore biomarkers of MS activity

CONTACTS AND LOCATIONS:
Overall Officials: Frank Valone, MD, Study Director — Bayhill Therapeutics
Locations (4):
- United States (2):
  - Barrow Neurology Clinics, Phoenix, Arizona
  - USC, LAC & USC Medical Center, Los Angeles, California
- Canada (2):
  - University of British Columbia, MS Research, Vancouver, British Columbia
  - Montreal Neurological Institute, Clinical Research Unit and MS clinic, Montreal, Quebec

REFERENCES:
- [Derived] Bar-Or A, Vollmer T, Antel J, Arnold DL, Bodner CA, Campagnolo D, Gianettoni J, Jalili F, Kachuck N, Lapierre Y, Niino M, Oger J, Price M, Rhodes S, Robinson WH, Shi FD, Utz PJ, Valone F, Weiner L, Steinman L, Garren H. Induction of antigen-specific tolerance in multiple sclerosis after immunization with DNA encoding myelin basic protein in a randomized, placebo-controlled phase 1/2 trial. Arch Neurol. 2007 Oct;64(10):1407-15. doi: 10.1001/archneur.64.10.nct70002. Epub 2007 Aug 13. PMID 17698695
- See also: Click here for more information about this study: BHT-3009-01 — http://www.webconferences.com/nihoba/ppt/633_RAC%20Vollmer%20present%206.8.04.pdf